CLINICAL TRIAL: NCT06836609
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of a Single Dose of ALN-CIDEB in Adult Participants With Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) and Two Doses of ALN-CIDEB in Adult Participants With Metabolic Dysfunction-Associated Steatohepatitis (MASH)
Brief Title: A Study to Evaluate ALN-CIDEB in Adult Participants With Metabolic Dysfunction-Associated Steatotic Liver Disease or With Metabolic Dysfunction-Associated Steatohepatitis (MASLD/MASH)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ALN-CIDEB-NASH-2486
Record Dates: First submitted 2025-02-14; First posted 2025-02-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Metabolic Dysfunction-Associated Steatohepatitis
Keywords: Obese; MASLD; MASH
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Part A: Sequential and Part B: Parallel
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Randomized per the protocol
  Interventions: Drug: ALN-CIDEB; Drug: Placebo
- Part B (Experimental): Randomized per the protocol
  Interventions: Drug: ALN-CIDEB; Drug: Placebo

INTERVENTIONS:
Drug: ALN-CIDEB — Administered per the protocol
Drug: Placebo — Administered per the protocol

SUMMARY:
This study is researching an experimental drug called ALN-CIDEB, also referred to as "study drug". The study is focused on participants with metabolic dysfunction-associated steatotic liver disease (MASLD) (Part A) and metabolic dysfunction-associated steatohepatitis (MASH) (Part B). MASLD and MASH are long-lasting liver conditions caused by having too much fat in the liver.

The aim of the study is to see how safe and tolerable the study drug is.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drug
* How the study drug works to change liver fat content
* How much study drug and study drug metabolites (byproducts of the body breaking down the study drug) are in the blood at different times

ELIGIBILITY:
Key Inclusion Criteria:

1. Part A: 18 to 55 years at Screening Visit 1 with MASLD, at Screening Visit 1 Part B: 18 to 65 years at Screening Visit 1 with a diagnosis of MASH, at Screening Visit 1
2. Body mass index (BMI) ≥30 kg/m2 and ≤40 kg/m2 at Screening Visit 1
3. Controlled-attenuation parameter (CAP) ≥270 dB/m by FibroScan during screening
4. Liver fat content ≥8.5% by MRI-PDFF during screening
5. If on anti-hypertensive and/or lipid lowering medications and/or glucose lowering medications, must be on generally stable dose(s) for at least 12 weeks prior to screening and no changes to the dose(s) are anticipated during the study
6. Part B: A diagnosis of MASH documented in the participant's medical history, or a clinical suspicion of MASH based on non-invasive biomarkers (eg, evidence of fatty liver on imaging and elevated liver enzymes) and clinical risk factors, including having a history of 2 or more elements of metabolic syndrome, as defined in the protocol
7. Part B: Screening percutaneous liver biopsy NAFLD Activity Score (NAS) ≥3 and fibrosis stage F0-F3, as defined in the protocol

Key Exclusion Criteria:

1. Known historical or current diagnosis of portal hypertension or cirrhosis based on clinical assessment, imaging, and/or liver biopsy
2. Known historical or current diagnosis of other forms of chronic liver disease, as defined in the protocol
3. Prior or current suspected or known drug-induced liver injury within 1 year prior to screening
4. History of liver transplant, current placement on a liver transplant list, or Model for End-stage Liver Disease (MELD) score >12
5. Contraindication to MRI examinations, such as persons with cardiac pacemaker and implants made of metal, severe claustrophobia, size restrictions, or other contraindications for MRI
6. Liver stiffness measurement, laboratory parameter assessment, estimated glomerular filtration rate (GFR), and evidence of uncontrolled hypertension, as defined in the protocol
7. Evidence of human immunodeficiency virus (HIV) infection, hepatitis B virus (HBV) infection, or hepatitis C virus (HCV) infection during screening, as described in the protocol
8. History of Type 1 Diabetes
9. Bariatric surgery within approximately 5 years prior to randomization or planned during the study period

NOTE: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | Up to 48 Weeks
Severity of TEAEs | Up to 48 Weeks

SECONDARY OUTCOMES:
Change in liver fat fraction by magnetic resonance imaging proton density fat fraction (MRI-PDFF) | Baseline up to 48 Weeks
Total concentration of ALN-CIDEB in plasma | Up to 48 Weeks
Total concentration of potential major metabolite(s) in plasma | Up to 48 Weeks
Urinary recovery of ALN-CIDEB as a proportion of the dose | Up to 36 Weeks
  Part A
Urinary recovery of potential major metabolite(s) as a proportion of the dose | Up to 36 Weeks
  Part A
Change in aspartate aminotransferase (AST) | Baseline up to 48 Weeks
Change in alanine aminotransferase (ALT) | Baseline up to 48 Weeks
Change in hepatic cell death-inducing DNA fragmentation factor alpha-like effector b (CIDEB) messenger RiboNucleic Acid (mRNA) level | Baseline up to 36 Weeks
  Part B

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Richmond Pharmacology Limited, London, Greater London
  - Parexel International Early Phase Clinical Unit, Harrow, London

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/